CLINICAL TRIAL: NCT00106132
Title: The Standard Care vs. Corticosteroid for Retinal Vein Occlusion (SCORE) Study
Brief Title: Steroid Injections vs. Standard Treatment for Macular Edema Due to Retinal Blood Vessel Blockage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050101; 05-EI-0101
Record Dates: First submitted 2005-03-19; First posted 2005-03-21 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-11

CONDITIONS: Retinal Vein Occlusion; Macular Edema, Cystoid; Macular Edema
Keywords: Macular Edema; Steroid; Fluorescein Angiogram; Ocular Coherence Tomography; Laser; Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide

SUMMARY:
This study will compare the safety and effectiveness of two treatments-injections of triamcinolone acetonide into the eye vs. standard laser therapy-for macular edema (swelling in the center of the retina) that is caused by blockage in a retinal blood vessel. Edema caused by blockage in a large vessel is called central retinal vein occlusion (CRVO). Edema caused by blockage in a smaller vein is called branch retinal vein occlusion (BRVO). Triamcinolone acetonide is a steroid drug that reduces swelling; the Food and Drug Administration has approved it for injection into joints and muscles to treat inflammatory conditions.

Patients 18 years of age and older with macular edema due to CRVO or BRVO of between 3 and 18 months' duration may be eligible for this study. Candidates are screened with a medical history, blood pressure measurement, and urine pregnancy test for women who can become pregnant. Screening also includes the following procedures:

* Eye examination to assess visual acuity and eye pressure, and to examine the cornea, lens, and retina. The pupils are dilated with drops for this examination.
* Fluorescein angiography to evaluate the eye's blood vessels. A yellow dye is injected into an arm vein and travels to the blood vessels in the eyes. Pictures of the retina are taken using a camera that flashes a blue light into the eye. The pictures show if any dye has leaked from the vessels into the retina, indicating possible blood vessel abnormality.
* Optical coherence tomography to measure retinal thickness. The eye is examined with a machine that produces cross-sectional pictures of the retina. The patient is seated in front of a machine and looks at a pattern of flashing and rotating red and green lights, first with one eye and then with the other.
* Fundus photography to help evaluate the status of the retina and changes that may occur in the future. Photographs of the retina are taken using a camera that flashes a bright light into the eye.

Participants are randomly assigned to receive triamcinolone injections or standard treatment. Triamcinolone is given in either a 1-mg or 4-mg dose. Standard treatment for CRVO and for BRVO with excessive blood in the retina is observation. Standard treatment for BRVO without excessive blood is laser therapy. Patients with BRVO who do not qualify for laser therapy when they enter the study may have it later if blood clears enough to permit treatment. The procedures for triamcinolone injections and laser therapy are as follows:

* Triamcinolone acetonide: The eye is numbed with anesthetic drops and the study drug is injected into the vitreous, the jelly-like substance located between the back of the lens and the retina. Patients apply antibiotic drops at home for 3 days following the procedure.
* Laser treatment: The eye is numbed with anesthetic drops and a special contact lens is placed on the eye during the laser beam application.

All patients are followed every 4 months for 3 years. Additional visits may be scheduled if needed. Patients who receive triamcinolone injections are also examined within 1 week of each injection and 1 month after each injection. At the 4-month visits patients undergo repeat eye examination and fundus photography. Optical coherence tomography is done at some visits, and fluorescein angiography is repeated at months 4, 12 and 24. Blood pressure is measured at months 12, 24 and 36. Patients may be retreated with triamcinolone injections or laser therapy as often as every 4 months, depending on their response to treatment.

DETAILED DESCRIPTION:
Macular edema is a major cause of vision loss in patients with central retinal vein occlusion (CRVO) and branch retinal vein occlusion (BRVO). Currently, there is no effective treatment for macular edema associated with CRVO. For macular edema associated with BRVO, grid laser photocoagulation may be an effective treatment, but many patients derive limited benefit from this treatment. Therefore, the development of new treatment modalities to treat macular edema caused by these two conditions is an important research goal. The Standard Care vs. COrticosteroid for REtinal Vein Occlusion (SCORE) Study will compare the efficacy and safety of standard care with intravitreal injection(s) of triamcinolone acetonide to treat macular edema associated with CRVO and BRVO.

The SCORE Study is designed as a multicenter, randomized, Phase III trial to compare the efficacy and safety of standard care versus triamcinolone acetonide injection(s) for the treatment of macular edema associated with CRVO and BRVO. In each of the two disease areas, 630 participants will be randomized in a 1:1:1 ratio to one of three groups: standard care, intravitreal triamcinolone 4 mg, or intravitreal triamcinolone 1 mg. For CRVO participants, standard care consists of observation of the macular edema. For BRVO participants, standard care consists of immediate grid laser photocoagulation for study eyes without a dense macular hemorrhage. For study eyes of BRVO participants with a dense macular hemorrhage, standard care is observation followed by grid laser photocoagulation if and when clearing of the hemorrhage permits grid laser photocoagulation. For all three groups, neovascular complications will be treated as necessary. Repeat treatments will be provided as clinically indicated based on protocol-specific guidelines. Participants will be followed for 3 years after randomization. The primary efficacy outcome of this study is improvement by 15 or more letters from baseline in best-corrected ETDRS visual acuity score at the 12-month visit. Secondary efficacy outcomes include change between baseline and each efficacy outcome assessment visit in best-corrected ETDRS visual acuity score, change in retinal thickness at the center of the macula and change in area of retinal thickening as assessed by stereoscopic color fundus photography, and change in retinal thickness and calculated retinal thickening as assessed by optical coherence tomography. Safety outcomes include injection-related adverse events such as infectious endophthalmitis, non-infectious endophthalmitis, retinal detachment, and vitreous hemorrhage and steroid-related adverse events, which include cataract and elevated intraocular pressure.

ELIGIBILITY:
INCLUSION CRITERIA:

General Inclusion Criteria:

* Ability and willingness to provide informed consent.
* Sex: Participants may be male or female.
* Age: 18 years or older

Ocular Inclusion Criteria (study eye):

A. Participants must have center-involved macular edema secondary to either CRVO or BRVO. Eyes may be enrolled if macular edema has been documented for at least 3 months and not longer than 18 months (by patient history or ophthalmologic diagnosis). The following definitions are used for the purposes of the SCORE Study:

* A CRVO is defined as an eye that has retinal hemorrhage or other biomicroscopic evidence of retinal vein occlusion (e.g. telangiectatic capillary bed) and a dilated venous system (or previously dilated venous system) in all 4 quadrants.
* A BRVO is defined as an eye that has retinal hemorrhage or other biomicroscopic evidence of retinal vein occlusion (e.g. telangiectatic capillary bed) and a dilated venous system (or previously dilated venous system) in 1 quadrant or less of retina drained by the affected vein.
* A hemiretinal vein occlusion (HRVO) is defined as an eye that has retinal hemorrhage or other biomicroscopic evidence of retinal vein occlusion (e.g. telangiectatic capillary bed) and a dilated venous system (or previously dilated venous system) in more than 1 quadrant but less than all 4 quadrants. Typically, a HRVO is a retinal vein occlusion that involves 2 altitudinal quadrants. For the purposes of the SCORE Study, eyes with HRVO will be treated as eyes with BRVO and analyzed with the BRVO group.

B. ETDRS visual acuity score of greater than or equal to 34 letters (approximately 20/200) and less than or equal to 73 letters (approximately 20/40) by the ETDRS visual acuity protocol at the screening visit.

C. Mean retinal thickness on two OCT measurements greater than or equal to 250 microns (central subfield) at the screening visit.

D. Media clarity, pupillary dilation and participant cooperation sufficient for adequate fundus photographs.

E. Stable visual acuity. This is defined as a less than 10 letter improvement in best-corrected ETDRS visual acuity score between the screening visit and the randomization visit. Those patients with a 10 or more letter improvement between the screening and randomization visits will be declared temporarily ineligible.

EXCLUSION CRITERIA:

General Exclusion Criteria:

Participants with any of the following conditions are ineligible:

A. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., chronic alcoholism or drug abuse, personality disorder or use of major tranquilizers indicating difficulty in long term follow-up, likelihood of survival of less than 3 years).

B. Participation in an investigational trial within 30 days of study entry that involved treatment with any drug that has not received regulatory approval at time of study entry.

C. History of allergy to any corticosteroid or component of the delivery vehicle.

D. Sitting systolic blood pressure greater than 180 mmHg or diastolic blood pressure greater than 110 mmHg at the screening visit. If the initial reading exceeds these values, a second reading may be taken two or more hours later; the patient may be included (if all other inclusion criteria are met) in the study if the second reading demonstrates a systolic blood pressure equal to or less than 180 mmHg and the diastolic blood pressure is 110 mmHg or less. If the blood pressure is brought to 180 mmHg systolic or less and 110 mmHg diastolic or less by antihypertensive treatment, the patient can become eligible.

E. The participant will be moving out of the area of the clinical center to an area not covered by another clinical center during the 3 years of the study.

F. History of systemic (e.g., oral, IV, IM, epidural, bursal) corticosteroids within 4 months prior to randomization or topical, rectal or inhaled corticosteroids in current use more than 2 times per week.

G. Positive urine pregnancy test: all women of childbearing potential (those who are pre-menopausal and not surgically sterilized) may participate only if they have a negative urine pregnancy test (at either the screening visit or randomization visit), if they do not intend to become pregnant during the timeframe of the study and if they agree to use at least one of the following birth control methods: hormonal therapy such as oral, implantable or injectable chemical contraceptives; mechanical therapy such as spermicide in conjunction with a barrier such as a condom or diaphragm; intrauterine device (IUD); or surgical sterilization of partner.

Ocular Exclusion Criteria (study eye):

A. Exam evidence of vitreoretinal interface disease (e.g. vitreomacular traction, epiretinal membrane), either on clinical examination or optical coherence tomography thought to be contributing to macular edema.

B. An eye that, in the investigator's opinion, would not benefit from resolution of macular edema such as eyes with foveal atrophy, dense pigmentary changes or dense subfoveal hard exudates.

C. Presence of an ocular condition that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., age-related macular degeneration, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, prior macula-off rhegmatogenous retinal detachment).

D. Presence of a substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more (i.e. a 20/40 cataract).

E. History of grid laser photocoagulation for macular edema.

F. History of intravitreal corticosteroid injection.

G. History of peribulbar or retrobulbar corticosteroid use for any reason within 6 months prior to randomization.

H. History of panretinal scatter photocoagulation (PRP) or sector laser photocoagulation within four months prior to randomization or anticipated within the next four months following randomization.

I. History of pars plana vitrectomy.

J. History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within 6 months prior to randomization or anticipated within the next 6 months following randomization.

K. History of YAG capsulotomy performed within 2 months prior to randomization.

L. IOP greater than or equal to 25 mm Hg.

M. Exam evidence of pseudoexfoliation.

N. History of steroid-induced IOP elevation that required IOP-lowering treatment.

O. History of open angle glaucoma (either primary open angle glaucoma or other cause of open angle glaucoma; note: prior angle closure glaucoma is not an exclusion).

* A history of ocular hypertension (or IOP greater than or equal to 22 mm Hg without a prior diagnosis of ocular hypertension) is not an exclusion as long as (1) IOP is less than 25 mm Hg, (2) the patient is using no more than one topical glaucoma medication, (3) the most recent visual field, performed within the last 12 months, is normal (if abnormalities are present on the visual field they must be attributable to the patient's macular disease), and (4) the optic nerve does not appear glaucomatous.
* Note: If IOP is 22 to less than 25 mm Hg, then the above criteria for ocular hypertension eligibility must be met.

P. History of herpetic ocular infection.

Q. History of ocular toxoplasmosis.

R. Aphakia.

S. Exam evidence of external ocular infection, including conjunctivitis, chalazion or significant blepharitis.

T. History of macular detachment.

U. Exam evidence of any diabetic retinopathy, defined as eyes of diabetic patients with more than one microaneurysm outside the area of the vein occlusion (inclusive of both eyes).

V. History of idiopathic central serous chorioretinopathy.

Fellow (Non-Study) Eye Criteria (the Fellow Eye Must Meet the Following):

A. ETDRS visual acuity score of greater than or equal to 19 letters (approximately 20/400)

B. No prior history of intravitreal corticosteroid injection.

C. IOP less than 25 mm Hg.

D. No exam evidence of pseudoexfoliation.

E. No history of steroid-induced IOP elevation that required IOP lowering treatment.

F. No history of open-angle glaucoma (either primary open-angle glaucoma or other cause of open-angle glaucoma; note: angle-closure glaucoma is not an exclusion).

* A history of ocular hypertension (or IOP greater than or equal to 22 mm Hg without a prior diagnosis of ocular hypertension) is not an exclusion as long as (1) IOP is less than 25 mm Hg, (2) the patient is using no more than one topical glaucoma medication, (3) the most recent visual field, performed within the last 12 months, is normal (if abnormalities are present on the visual field they must be attributable to the patient's macular disease), and (4) the optic nerve does not appear glaucomatous.
* Note: If the IOP is 22 to less than 25 mm Hg, then the above criteria for ocular hypertension must be met

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1260
Dates: Start 2005-03; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Patz A. Argon laser photocoagulation for macular edema in branch vein occlusion. Am J Ophthalmol. 1984 Sep 15;98(3):374-5. doi: 10.1016/0002-9394(84)90331-3. No abstract available. PMID 6540993
- [Background] Opremcak EM, Bruce RA. Surgical decompression of branch retinal vein occlusion via arteriovenous crossing sheathotomy: a prospective review of 15 cases. Retina. 1999;19(1):1-5. doi: 10.1097/00006982-199901000-00001. PMID 10048366
- [Background] Baseline and early natural history report. The Central Vein Occlusion Study. Arch Ophthalmol. 1993 Aug;111(8):1087-95. doi: 10.1001/archopht.1993.01090080083022. PMID 7688950